CLINICAL TRIAL: NCT05764317
Title: DescripTion of the Effectiveness, Safety, Tolerability and Adherence to Amlodipine/atoRvastatin/Perindopril sinGle Pill Combination trEatmenT in Patients With Arterial Hypertension and Dyslipidemia in the Daily Clinical Practice. (TARGET)
Brief Title: Description of the Effectiveness, Safety, Tolerability and Adherence to Amlodipine/Atorvastatin/Perindopril Single Pill Combination Treatment in Patients With Arterial Hypertension and Dyslipidemia (TARGET)
Acronym: TARGET
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05153-070-RUS
Record Dates: First submitted 2023-02-09; First posted 2023-03-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Arterial Hypertension; HTN
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Atorvastatin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Amlodipine 5 mg + atorvastatin 10 mg + perindopril arginine 5 mg — a triple fixed combination of atorvastatin, perindopril and amlodipinedose combinations, was in a 3-month in accordance to the instruction for medical use approved in the Russian Federation
Drug: Amlodipine 5 mg + atorvastatin 20 mg + perindopril arginine 5 mg — a triple fixed combination of atorvastatin, perindopril and amlodipinedose combinations, was in a 3-month in accordance to the instruction for medical use approved in the Russian Federation
Drug: Amlodipine 5 mg + atorvastatin 20 mg + perindopril arginine 10 mg — a triple fixed combination of atorvastatin, perindopril and amlodipinedose combinations, was in a 3-month in accordance to the instruction for medical use approved in the Russian Federation

SUMMARY:
This is a multi-centre, observational, ambispective study, which will retrospectively and prospectively collect clinical and socio-demographic data from medical records of patients with HTN and dyslipidemia initiated with SPC of amlodipine/atorvastatin/perindopril in real clinical settings.

A total of 80 general practitioners and outpatient cardiologists will participate in this non-interventional study 400 patients should be included in the study.

DETAILED DESCRIPTION:
Treatment with the studied drug:

* Amlodipine 5 mg + atorvastatin 10 mg + perindopril arginine 5 mg
* Amlodipine 5 mg + atorvastatin 20 mg + perindopril arginine 5 mg
* Amlodipine 5 mg + atorvastatin 20 mg + perindopril arginine 10 mg This is non-interventional study that is observational by its nature. Therefore there will be no any assignments of subjects to a particular therapeutic strategies defined by this protocol. Decision to treat a patient with SPC of amlodipine/ atorvastatin/ perindopril should be at the descretion of a treating investigator and made in accordance to local standards and protocols.

ELIGIBILITY:
Inclusion Criteria:

* Obtained signed informed consent from the patient
* Patients of 18 years and older and younger than 80 years.
* Start of the treatment with SPC of amlodipine/atorvastatin/perindopril within 1 month from the Index date in accordance with the indication in Russian SmPC.
* Presence of the parameters of interest* in the medical records dated with the nearest to the start of SPC amlodipine/atorvastatin/perindopril treatment date.

  * Parameters of interest include measured at rest office BP and LDL-C.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide a signed informed consent form;
* Any contraindication to the treatment with the SPC of amlodipine/atorvastatin/perindopril according to its' approved instruction for medical use in the Russian Federation;
* Concomitant use of any other ACE inhibitors, CCBs, ARBs and statins.
* Supposed low treatment adherence to the assigned SPC and the risk for poor collaboration between the patient and the investigator during the study;
* Any severe, decompensated or unstable somatic diseases or states that according to investigator discretion are life-threatening or worsen the prognosis for the patient: myocardial infarction in the past 3 months, unstable angina, current decompensation of diabetes mellitus, autoimmune or oncological diseases, severe cardiac arrhythmia, gastrointestinal disorders affecting absorbtion, severe hepatic diseases, pancreatic diseases, severe allergic reactions, connective tissue diseases etc;
* Secondary arterial hypertension;
* Alcohol or any drug abuse;
* Surgical intervention on heart or coronary vessels (i.e., heart valve(s) replacement, stent implantation or CABG), or any non-cardiological serious surgical intervention that are planned within next 3 months and may require withdrawal or changes in current therapy;
* Glomerular filtration rate less than 60 ml/min/1,72m2;
* Participating in any other clinical trial currently or during 30 days period before informed consent was signed.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with HTN and dyslipidemia who had been initiated with SPC amlodipine/atorvastatin/perindopril within one month before the inclusion
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
To describe antihypertensive effectiveness of a triple single-pill combination of amlodipine, atorvastatin and perindopril at 12 weeks in patients with arterial hypertension (HTN) and dyslipidemia in the daily clinical practice. | 12 weeks
  Mean change from baseline in SBP (systolic blood pressure) and DBP (diastolic blood pressure) assessed at week 12 of the observational period.
To describe hypolipidaemic effectiveness of a triple single-pill combination of amlodipine, atorvastatin and perindopril at 12 weeks in patients with arterial hypertension (HTN) and dyslipidemia in the daily clinical practice. | 12 weeks
  Mean change from baseline in LDL-C ( low density lipoprotein cholesterol) assessed at week 12 of the observational period

SECONDARY OUTCOMES:
To determine the proportion of patients who reached systolic (SBP) and diastolic blood pressure (DBP) target goals at weeks 4 and 12 of the observation period respectively. | 12 weeks
To determine the proportion of patients who reached LDL-C target goals at week 12 of the observation period. | 12 weeks
To evaluate the quality of life of patients at visit 1 (V1) and visit 2 (V2) as compared to visit 0 (V0) respectively | 12 weeks
  Mean change from V0 in scores of the SF-36 questionnaire assessed at V1 and V2;
To evaluate the adherence to treatment with the fixed dose combination of amlodipine/atorvastatin/perindopril in patients included into the study at V1 and V2 as compared to V0 | 12 weeks
  Proportion of patients with high, moderate and low adherence to the treatment with SPC (single pill combination) of amlodipine/atorvastatin/perindopril at V1 as compared to V0 via medication adherence scale; Proportion of patients with high, moderate and low adherence to the treatment with SPC of amlodipine/atorvastatin/perindopril at V2 as compared to V0 via medication adherence scale;
To evaluate predictors of reaching BP target goals in the study population | 12 weeks
  Proportion of patients achieving target BP levels depending on baseline SBP and DBP;
To evaluate predictors of reaching LDL-C target goals in the study population | 12 weeks
  Proportion of patients achieving target levels LDL C depending on baseline LDL-C level.

CONTACTS AND LOCATIONS:
Locations (1):
- Servier, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT05764317/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT05764317/ICF_001.pdf